CLINICAL TRIAL: NCT01005225
Title: Genetic Investigation of Solid Tumors Cohort
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: HSC# 004835
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer; Colon Cancer
Keywords: Solid tumor; prostate cancer; colon cancer
MeSH Terms: conditions — Prostatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Approximately 19.5 milliliters (mls) of blood will be collected in (2 x 8.5 ml) PAXgene DNA tubes and (1 x 2.5 ml) PAXgene RNA tube.
  Solid tumor and/or benign hyperplasia samples will be collected from the participants during surgery scheduled for standard medical care.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Solid tumors: Participants 18 years of age or older who have been diagnosed with a solid tumor or benign hyperplasia that needs surgical removal will be included in this study.

SUMMARY:
The objective of this study is to obtain blood samples, solid tumor and/or benign hyperplasia samples to learn more about genetic differences that are linked to the formation of solid tumors.

DETAILED DESCRIPTION:
Recent studies in human genetics have discovered several intervals in the human genome containing inherited variants that are statistically associated with the propensity to develop solid tumors. Even though it has been firmly established that if an individual carries these DNA variants they have an increased chance of developing a solid tumor the underlying biological mechanisms for most of these associations are largely unknown.

In addition to inherited DNA variants that are associated with the development of solid tumors it is well established that during the development and growth of solid tumors the DNA in these cancer cells undergo somatic changes (mutations). These somatic DNA changes have been studied over the past decade and frequently are specific chromosomal translocations and amplifications associated with the development of particular solid tumors. In some instances, examining the chromosomal translocation and amplification has lead to the discovery of proteins contributing to solid tumor pathology.

the human 8q24 interval that has strong genetic associations with solid tumor development has also been noted as frequently amplified in solid tumors and serves as a predictor of poor survival in prostate cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Eligible to have their blood drawn
3. Be reliable, cooperative and willing to comply with all protocol-specified procedures
4. Able to understand and grant informed consent
5. Diagnosis of a solid tumor

Exclusion Criteria:

1. Has a significant chronic medical condition which would potentially confound interpretation of the individual's phenotype.
2. Treatment with any investigational agents or devices within thirty days preceding enrollment in the study.
3. Been administered or taken any CNS sedatives or depressants in the 12 hours prior to informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic, physician referral
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Solid tumor biological insights | Study completion
  Obtain blood samples, solid tumor and/or benign hyperplasia samples, and in some instances normal tissue in order to gain biological insights into cancer (solid tumors) through population genetics and genomics.

CONTACTS AND LOCATIONS:
Overall Officials: James Mason, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Health, San Diego, California, United States